CLINICAL TRIAL: NCT03361644
Title: The Role of High Intensity Interval Training in the Treatment of Adolescent Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20010365; R21HD090448 (NIH)
Record Dates: First submitted 2017-11-17; First posted 2017-12-05 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pediatric Obesity; Adolescent Obesity; Weight Loss
MeSH Terms: conditions — Pediatric Obesity; Weight Loss | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 2x3 repeated-measures randomized control trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Interval Training (Experimental): Brief periods of vigorous physical activity separated by short periods of rest.
  Interventions: Behavioral: High-Intensity Interval Training
- Moderate-Intensity Continuous Training (Active Comparator): Physical activity at a sustained moderate heart rate.
  Interventions: Behavioral: Moderate-Intensity Continuous Training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Participants assigned to HIIT will participate in treadmill exercise in intervals consisting of 1 minute intervals of challenging intensities with recovery periods in between, gradually increasing the number of intervals over the course of the study.
  Arms: High-Intensity Interval Training
Behavioral: Moderate-Intensity Continuous Training — Participants assigned to CMIT will participate in constant moderate intensity treadmill exercise, gradually increasing the duration of the exercise over the course of the study.
  Arms: Moderate-Intensity Continuous Training

SUMMARY:
The study will compare the effects of High Intensity Interval Training (HIIT) with Moderate Intensity Continuous Training (CMIT) as part of a lifestyle intervention program on BMI change in adolescents age 12-16 with obesity.

DETAILED DESCRIPTION:
Adolescents will be randomized to a 12-week lifestyle intervention including behavioral and dietary interventions, and one of two exercise training conditions, HIIT or CMIT). Adolescents in the HIIT treatment will participate in treadmill exercise in 1-minute intervals of challenging intensities with recovery periods in between, gradually increasing the number of intervals over the course of the study. Adolescents in the CMIT treatment will participate in a constant moderate intensity treadmill exercise, gradually increasing the duration of the exercise over the course of the study.

Both parents and teens will have height and weight measurements taken, complete behavior questionnaires and wear an activity monitor for one week at baseline, 12 weeks and 16 weeks.

Adolescents will have a physical exam by a study medical provider before starting the intervention. Adolescents will also have blood work, an oral glucose tolerance test, an electrocardiogram, body composition measurements and a maximal graded exercise test done at baseline, and again at one or more time points. Adolescents will also complete a detailed food log at those time points.

Adolescents will exercise at the study gym 3 evenings a week for 12 weeks. On one of those evenings teens will also attend a 60-minute individual behavioral weight management session. Nine of these are with a behavior coach, and 3 with a dietitian. Parents will also attend one introductory session with the behavior coach, join the teen for the 3 sessions with the dietitian, and review adolescent individual goals and identify parent support goals at the end of each behavior session.

ELIGIBILITY:
Inclusion Criteria:

* Age of 12 to 16 years with obesity (BMI ≥95% percentile for age and gender according to the CDC Growth Charts).
* Have a parent (or legal guardian) who is willing to provide basic demographic information, complete required surveys, and attend portions of the weekly adolescent-focused behavioral weight management sessions.
* Participating parent must reside with the adolescent within a 30-mile distance of the study site.

Exclusion Criteria:

* Non-English speaking;
* Weight >300 lbs;
* Medical condition(s) that may be associated with unintentional weight change (e.g., hypothalamic injury, Prader-Willi, untreated thyroid disease or malignancy);
* Diabetes mellitus diagnosed by history or a fasting glucose ≥126 mg/dl (subjects with glucose intolerance or "prediabetes" will eligible for study participation);
* Use of insulin sensitizing agents (e.g. metformin), antihypertensive medications, medications for treatment of hyperlipidemia, oral contraceptives, oral glucocorticoids, atypical antipsychotics, weight loss medications, or an investigational medication within 3 months of study participation;
* Medical condition(s) that may be negatively impacted by high-intensity exercise training;
* Psychiatric, cognitive, developmental or physical conditions that would impair the adolescent's ability to complete assessments, participate in behavioral weight management sessions, or conduct physical activity;
* Reports of compensatory behaviors (i.e., vomiting, laxative abuse, excessive exercise) in the past 3 months;
* Current pregnancy or plan to become pregnant during study period;
* Previous participation in the TEENS study at Virginia Commonwealth University;
* Current participation in another weight loss program; or
* Personal history of weight loss surgery;

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 12 weeks
  The two training methods will be compared for how they impact participants' fitness levels as assessed during a graded exercise tolerance test.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | 12 weeks
  The two training methods will be compared for changes in participants' BMI in kg/m2
Change in Blood Lipid Levels | 12 weeks
  The two training methods will be compared for changes in fasting lipid levels.
Change in Body Composition | 12 weeks
  The two training methods will be compared for differences in changes of percent body fat.
Participant Attendance | 12 weeks
  The two training methods will be compared for differences in rates of participant attendance at intervention sessions.
Achievement of Heart Rate Goals. | 12 weeks
  The two training methods will be compared for differences in rates of achievement of heart rate goals during exercise training sessions.
Acceptability of exercise | 12 weeks
  The two training methods will be compared for differences in participants' reported enjoyment of the exercise session.
Feasibility of Exercise | 12 weeks
  The two training methods will be compared for differences in participants' confidence in being able ability to continue to participate in the assigned type of exercise.
Maintenance of lifestyle changes | 16 weeks
  The two training methods will be compared for participants' frequency of participation in physical activity 1 month after completion of the intervention.
Weight loss maintenance | 16 weeks.
  The two training methods will be compared for changes in BMI 1 month after completion of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Edmond P Wickham, MD, Principal Investigator — VCU Departments of Pediatrics and Internal Medicine
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03361644/ICF_000.pdf